CLINICAL TRIAL: NCT05222243
Title: Evaluation of Calcium Hydroxide Paste, Mineral Trioxide Aggregate and Formocresol as A Direct Pulp Capping in Primary Molars. Randomized Controlled Clinical Trial
Brief Title: DPC in Primary Molars.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05030718
Record Dates: First submitted 2021-12-08; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2018-07

CONDITIONS: Direct Pulp Capping in Primary Teeth
MeSH Terms: interventions — Calcium Hydroxide; Pemetrexed; formocresol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calcium Hydroxide (CH) (Active Comparator): Calcium Hydroxide is the gold standard for direct pulp capping depends on regeneration
  Interventions: Drug: Direct pulp capping with calcium hydroxide
- MTA (Experimental): Mineral trioxide aggregate used for pulp regeneration
  Interventions: Drug: Direct pulp capping with MTA
- Formocresol (FC) (Experimental): composed of formaldehyde, cresol, glycerin and water used for fixation of pulp tissue
  Interventions: Drug: Direct pulp capping with Formocresol

INTERVENTIONS:
Drug: Direct pulp capping with calcium hydroxide — Capping exposed dental pulps during cavity preparation in primary teeth with calcium hydroxide
  Arms: Calcium Hydroxide (CH)
Drug: Direct pulp capping with MTA — Capping exposed dental pulps during cavity preparation in primary teeth with MTA
  Arms: MTA
Drug: Direct pulp capping with Formocresol — Capping exposed dental pulps during cavity preparation in primary teeth with zinc oxide eugenol after medication with formocresol
  Arms: Formocresol (FC)

SUMMARY:
To evaluate clinical and radiographical outcomes of direct pulp capping using calcium hydroxide (CH), mineral trioxide aggregate (MTA), and premedicated direct pulp capping (PDPC) with formocresol (FC) in primary teeth.

DETAILED DESCRIPTION:
The pulp is imperiled by many environmental impacts. Caries, trauma, restorations, and mechanical injury during cleaning, all are possible aggressions that may injury the pulp tissue. When lesion disrupt enamel barrier, dentin can be degraded by Gram-positive bacteria, such as actinomyces, lactobacilli, and streptococci, that largely dominate the microflora of carious lesion. Pulp response differs according to the degree of the insult. The inflammatory reaction can cause permanent damage or be followed by repair, as the pulp cells have the ability to differentiate into odontoblasts forming dentin matrix facilitating wound healing.

Calcium hydroxide was introduced to the dental practice in the 1920s, and early clinical studies using it in direct pulp capping showed an 80-90 percent success rate.Recent studies with longer follow-up periods suggest lower success rates for it.Calcium hydroxide was used in many forms alone and mixed with other materials for many applications in the dental profession. For direct pulp capping calcium hydroxide powder and aqueous paste were used at first then premixed and cement-based types were developed.

Mineral trioxide aggregate (MTA) was introduced to the dental practice in the 1990s as a root-end filling material. MTA is used as a gold standard in endodontics and has a variety of applications such as root-end filling, apexification, root and truck perforations, apexogenesis, pulp capping in permanent and primary teeth, and dressing for pulpotomy in primary teeth. It is mainly composed of tricalcium silicate, tricalcium aluminate, dicalcium silicate, bismuth oxide, and calcium sulfate dehydrate.

Several studies have shown the efficacy of direct pulp capping using calcium hydroxide and MTA in permanent teeth. However, its use in primary teeth is controversial and few studies are available regarding that subject. Formocresol is not known to be used in direct pulp capping techniques, however, its high clinical success in pulpotomy techniques for primary teeth promoted the investigation of its possible use as direct capping medicament. In addition, there are not enough collected clinical and histological data about direct capping in primary teeth to assess the true success of treatment. Accordingly, the study was directed to evaluate the histological and clinical success of different materials in direct pulp capping for primary teeth.

ELIGIBILITY:
Inclusion Criteria:

1. Absence of chronic systemic disease and any type of medical treatment or continues use of any medication.
2. Absence of drug allergies, anesthetics, and environmental allergies.
3. Cooperative patients.
4. Restorable teeth with deep decay lesions.
5. Teeth with signs of reversible pulpitis; no spontaneous pain; and absence of edema, pain, fistula, pathological mobility, and sensitivity to percussion.
6. True pinpoint exposure (small exposure surrounded by sound dentin with normal bleeding easily controlled)
7. Teeth with no pathological root resorption, periradicular or furcal radiolucency.
8. Teeth with less than one-third physiological root resorption (no resorption or one-fourth resorption of the root).

Exclusion Criteria:

* otherwise

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Radiolucency of the periapical or furcation area | 12 months
  measuring tool is x-ray

SECONDARY OUTCOMES:
Pathological internal or external root resorption | 12 months
  measuring tool is x-ray
Widening of the periodontal space | 12 months
  measuring tool is x-ray
Calcification of the pulp canal | 12 months
  measuring tool is x-ray
Spontaneous pain | 12 months
  numeric rating scale (presence or abscence of pain) 0 is best result 10 is the worst
Sensitivity on percussion and palpation | 12 months
  methods of tapping on surface in clinical examination
Presence or absence of fistula | 12 months
  visual inspection
Pathological mobility | 12 months
  mobility is graded clinically by applying pressure with ends of two metal instruments

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR